CLINICAL TRIAL: NCT00476463
Title: Virological and Clinical Anti-HBV Efficacy of Tenofovir and Emtricitabine in Antiretroviral Naive Patients With HIV/HBV Co-infection
Brief Title: Efficacy of Tenofovir and Emtricitabine in ARV-naive Patients With HIV/HBV Co-infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Gilead Sciences (Industry); Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 023
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B Virus; HIV Infections
Keywords: TDF+FTC; FTC; HIV/HBV; TDF compared to TDF+FTC in HIV/HBV; Treatment Naive
MeSH Terms: conditions — Hepatitis B; HIV Infections | interventions — Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): AZT+FTC+EFV
  Interventions: Drug: Emtricitabine
- 2 (Active Comparator): TDF+FTC+EFV
  Interventions: Drug: Emtricitabine

INTERVENTIONS:
Drug: Emtricitabine — Emtricitabine 200 mg OD + Zidovudine 300 mg BID + EFV OD compared to TDF + FTC + EFV

SUMMARY:
Combination therapy with anti-HBV activity may both increase HBV suppression rates and reduce emergence of resistant strains. Several new therapeutic agents are currently in development, however combination therapy trials in the HBV-infected population have only recently commenced. No such trials have been undertaken in the HIV/HBV co-infected population.

DETAILED DESCRIPTION:
The primary study objective is to compare HBV DNA suppression to levels below the limit of detection (<400 copies/ml) by week 48 in each treatment group. Virological and clinical anti-HBV efficacy of tenofovir and emtricitabine in antiretroviral naive patients with HIV/HBV co-infection.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Documented HIV infection (positive serology for HIV-1 and detectable HIV-1 RNA)
* Age 18 - 70 years
* HBV DNA > 106 copies/ml
* HBsAg positive for > 6 months

In case documented duration of HBsAg seropositive is less than 6 months (this situation is most likely to occur in patients newly presenting to the HIV-outpatient clinic) the patient is eligible if the patient is:

1. HBsAg positive and
2. HBc core IgM antibody negative and
3. the liver biopsy gives evidence for a chronic active hepatitis. Thus making it likely that this patient has acquired the HBV infection more than 6 months ago.

   * ALT < 10 x ULN
   * Creatinine <= 2.0mg/dl
   * Platelet count >= 50,000/mm3
   * HIV-1 therapy naive
   * No prior exposure to anti-HBV agents (LAM, adefovir, TDF) although prior IFN treatment allowed

Exclusion Criteria:

* HCV-RNA positive or Anti-HAV IgM positive
* Acute hepatitis (serum ALT > 1000 U/L)
* Prior LAM, TDF, or ADV therapy
* Active opportunistic infection
* Other causes of chronic liver disease identified ( autoimmune hepatitis, haemochromatosis, Wilsons disease, alfa-1-antitrypsin deficiency)
* Concurrent malignancy requiring cytotoxic chemotherapy
* Decompensated or Child's C cirrhosis
* Alfa-fetoprotein (AFP) > 3X ULN (unless negative CT scan or MRI within 3 months of entry date)
* Pregnancy or lactation
* Any other condition which in the opinion of the investigator might interfere with compliance or outcome of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
HBV DNA suppression to levels below the limit of detection (<400 copies/ml) | week 48

SECONDARY OUTCOMES:
HBV suppression as measured by comparison of AUC measurements at 12 and 24 weeks | 12 and 24 weeks
Proportion of patients with undetectable HBV DNA in serum at 12 and 24 weeks | 12 and 24 weeks
Rate of HBeAg and HBsAg seroconversion at 12, 24 and 48 weeks. | 12, 24 and 48 weeks
Rate of emergence of LAM-resistant HBV genotypes at 48 weeks. | 48 weeks
Rate of hepatic cytolysis (ALT level > 5x ULN). | 48 weeks
Change from baseline in ALT levels and time to ALT normalization. | 48 weeks
Suppression of plasma HIV-RNA (< 50 copies/ml) through 48 weeks. | 48 weeks
Changes in CD4+ /CD8+ cell counts through 48 weeks | 48 weeks
Toxicity | 48 weeks
Assessment of effect of therapy on histological changes in the liver and effect on ccc-HBV-DNA | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — HIV-NAT Thai Red Cross AIDS Research Center
Locations (1):
- HIV-NAT Thai Red Cross AIDS Research Center, Bangkok, Thailand

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org